CLINICAL TRIAL: NCT03441542
Title: A Randomized Study of the Effectiveness of Patient Registry Directed Patient Navigation in Improving Attainment of Hepatitis C Virus (HCV) Care Among Patients Using Opioid Substitution Therapy and Patients Who Currently Inject Drugs
Brief Title: Registry-based HCV Care Cascade Navigation at Atlanta's Grady Memorial Hospital
Acronym: EZ-C
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment. Reasons for low enrollment were low eligibility, and difficulty contacting patients.
Sponsor: National Opinion Research Center (Other)
Collaborators: Grady Health System (Other); Merck Sharp & Dohme LLC (Industry); Emory University (Other)
Responsible Party: Principal Investigator, Dr. David Rein, Program Area Director, Public Health, National Opinion Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 8223
Record Dates: First submitted 2018-02-09; First posted 2018-02-22 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Hepatitis C
Keywords: Care cascade; Patient navigation services; Injection drug users; Opioid substitution therapy
MeSH Terms: conditions — Hepatitis C | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Data-assisted Case Navigation (Experimental): Patients are recruited and consented into the study by the patient navigator after which the navigator provides assistance with scheduling, reminders, and transportation. The navigator is also charged with responding to patient questions, and monitoring and documenting if and when patients achieve HCV care milestones. Each month, the project will update the Grady Liver Clinic HCV patient registry, to generate information about the patient's HCV care progress and use this information to develop instructions sheets regarding the expected care milestones to be achieved that month for each patient. During the month, the navigator will participate in project meetings and report on milestone achievement and barriers for patients assigned to the experimental arm of the study.
  Interventions: Behavioral: Data-assisted Case Navigation
- Standard of Care (Active Comparator): Patients are recruited and consented into the study by the patient navigator at which time they will be reminded of their infection, consequences of untreated disease, and the availability of study sponsored antiviral treatment should they seek it. Patients will not be subsequently contacted by the study. Patients who seek treatment without patient navigation services will receive the same study provided HCV pre-treatment care and study provided treatment drugs when indicated. Self-referral to care and antiviral therapy when indicated are known to be effective in curing HCV among some patients, this arm is classified as an active comparator.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Data-assisted Case Navigation — The researchers will develop a monthly task list for the patient navigator with patient by patient care cascade and treatment milestones that need to be accomplished per patient in the case group. The researchers will deliver the spreadsheet and the task list to the Grady Liver Clinic Director who will use it to direct and supervise the activities of the patient navigator.
  Patient navigators will be responsible for reaching out to patients in only the intervention arm about their next step in the HCV care cascade.
  Arms: Data-assisted Case Navigation
Behavioral: Standard of Care — Patients will be recruited into the study by the patient navigator, be provided information about HCV infection, and will be informed that treatment is freely available should they seek it. Patients will also be provided contact and address information for the treatment clinic.
  Arms: Standard of Care

SUMMARY:
This study seeks to implement and evaluate a data-driven case navigation system for hepatitis C virus (HCV) treatment among persons who are either actively injecting drugs or who are receiving opioid substitution therapy (OST). The study will use data from a previously developed patient registry system to identify patients for study recruitment, and use monthly updates of registry data to organize and direct patient navigation services for those individuals assigned to the treatment group. Patients assigned to the control group will also be eligible to receive HCV treatment, but will otherwise receive usual care.

This study has a parallel, randomized unblinded, case/control design in which eligible patients are assigned at baseline to either a registry-directed patient navigation system (case) or to usual care (control), characterized in terms of demographic and sub-population variables, and then compared after 12 months on two categories of outcomes; (1) attainment of care cascade milestones; and (2) treatment initiation, adherence, and virologic response. The study is designed and powered to answer two primary hypotheses (H1 & H2):

* H1: As compared to those randomized to usual care (control), those randomized to the registry directed patient navigation arm (case) will be more likely to complete all pretreatment HCV care milestones as defined by a higher proportion completing all four pre-treatment care cascade outcomes.
* H2: As compared to the control group, a significantly higher proportion of those randomized to the case group will achieve a sustained viral response.

DETAILED DESCRIPTION:
EZ-C's purpose is to determine the effectiveness of patient navigation services during treatment of hepatitis C compared to usual care among opioid substitution therapy (OST) and active injecting drug use (IDU) individuals.

To recruit OST and active IDU patients, customized queries will be created to identify pharmaceutical (methadone, buprenorphine, buprenorphine/naltrexone, naloxone) and diagnostic (ICD-10 codes for heroin poisoning, history of heroin abuse, long term current use of opiate analgesic, opioid dependence, and potentially others) indicators of OST or active injecting drug use. These codes will be implemented into the Grady HCV registry to flag and identify OST or possible active injecting drug use individuals that are HCV positive at Grady Health Systems.

Recruitment will consist of an initial letter describing the study and informing patients of their possible eligibility as well as informed consent documentation. This letter will be followed by up to three phone calls per patient from the patient navigator until a full sample of OST and active injecting drug users have been recruited. Once enrolled, patients will be randomly assigned into either the control or intervention group. Although there is no compensation for participating in the study, all patients that are recruited will receive treatment at no cost.

Once the study begins enrolling, the researchers will create spreadsheet reports of patients in the intervention group (those who are receiving patient navigation services) containing their HCV care information, such as antibody results, viral load test results and prescription refill information. Based on this spreadsheet, the researchers will develop a monthly task list for the patient navigator with patient by patient care cascade and treatment milestones that need to be accomplished per patient in the intervention group. The researchers will then deliver the spreadsheet and the task list to the Grady Liver Clinic Director who will use it to direct and supervise the activities of the patient navigator. The patient navigator will actively engage with those in the intervention group throughout the study and send reminders of their next steps in the treatment process/care cascade. The patient navigator will not engage with those in the control group as they will receive only usual care.

The intervention will last 12 months for each patient in both the case and control groups. After collecting data for the 80 patients at the end of the study, the researchers will analyze the data to determine the effectiveness of patient navigation services compared to those receiving usual care among IDU and OST individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is antibody positivity for HCV, defined as;

   * Patients identified in the Grady Memorial Hospital Hepatitis C registry who have tested antibody positive for HCV and have not received additional RNA confirmatory or genotype testing; or
   * Patients who tested antibody positive for HCV through Grady Liver Clinics allied community-based testing organizations.
2. Patient is a member of one of two sub-population groups of interest, people on opioid substitution therapy (OST) or people who currently inject drugs, defined as;

   * A pharmaceutical or diagnostic indicator of OST or morbidity resulting from injecting drug use identified in the patient's electronic health record (EHR), or
   * Referral for HCV care from an Atlanta area syringe exchange program
3. Eligible for treatment. To be eligible for treatment, patients must

   * Meet the above criteria,
   * Complete care milestones of viral load/RNA confirmation, viral genotyping, clinical evaluation, and non-invasive fibrosis stages;
   * Exhibit a detectable viral load, and an HCV genotypes of 1 or 4
   * Note: Enrolled patients infected with genotypes other than 1 or 4 will be treated according to usual care practices of the Grady Liver Clinic.

Exclusion criteria. Patients who meet criteria 1 and 2 will be excluded from the study if

* They have already received confirmatory RNA or genotype testing
* Have been offered treatment by the Grady Liver Clinic and refused
* Have a comorbidity that the Grady Liver Clinic determines would contraindicate treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Completion of HCV care milestones in HCV cure cascade | Within 6 months of enrollment
  Variable indicating which step in the cure cascade patient last completed

OTHER OUTCOMES:
Achievement of HCV sustained viral response (SVR) | Within 12 months of enrollment
  Dichotomous (yes/no) variable of achieving SVR

CONTACTS AND LOCATIONS:
Overall Officials: David Rein, Ph.D., Principal Investigator — NORC at the University of Chicago
Locations (1):
- Grady Health System, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No